CLINICAL TRIAL: NCT00410202
Title: A Comparative Study of Entecavir vs. Adefovir Plus Lamivudine vs Combination Entecavir Plus Adefovir in Lamivudine-resistant Chronic Hepatitis B Subjects: The DEFINE Study
Brief Title: Entecavir Plus Adefovir Combination Therapy Versus Entecavir Monotherapy vs Therapy With Adefovir Plus Lamivudine for Chronic Hepatitis B Infected Subjects With Lamivudine-resistant Virus
Acronym: DEFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-111
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; adefovir; adefovir dipivoxil; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Entecavir (Active Comparator): With the option of adding tenofovir at week 48. (This does not apply to Korea)
  Interventions: Drug: Entecavir; Drug: Tenofovir
- Adefovir + Lamivudine (Active Comparator)
  Interventions: Drug: Adefovir; Drug: Lamivudine
- Entecavir + Adefovir (Active Comparator)
  Interventions: Drug: Entecavir; Drug: Adefovir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 1mg, once daily, 100 weeks
  Other Names: Baraclude; BMS-200475
  Arms: Entecavir; Entecavir + Adefovir
Drug: Tenofovir — Tablets, Oral, 300 mg, once daily
  Other Names: Viread
  Arms: Entecavir
Drug: Adefovir — Tablets, Oral, 10mg, once daily, 100 weeks
  Other Names: Hepsera
  Arms: Adefovir + Lamivudine; Entecavir + Adefovir
Drug: Lamivudine — Tablets, Oral, 100mg, once daily, 100 weeks
  Other Names: Epivir
  Arms: Adefovir + Lamivudine

SUMMARY:
The purpose of this study is to evaluate the effectiveness of entecavir plus adefovir combination therapy versus entecavir monotherapy or therapy with adefovir plus lamivudine

ELIGIBILITY:
Inclusion Criteria:

* Evidence of lamivudine (LVD) resistance
* Subjects must have a history of previous LVD treatment at screening, and must have evidence of at least 1 LVD resistance substitution (valine, isoleucine, or serine) at reverse transcriptase codon 204 (M204V/I/S)
* Nucleoside- and nucleotide-naive, except for LVD, and had chronic hepatitis B (HBV) infection
* Compensated liver function and must have met ALL of the following criteria:International normalization ratio (INR) ≤ 1.5; Serum albumin ≥ 3 g/dL (≥ 30 g/L); Serum total bilirubin ≤ 2.5 mg/dL (≤ 42.75 μmol/L)
* HBV DNA > 1.72 x 10*4* IU/mL (approximately 10*5* copies/mL)
* Documentation of hepatitis B e antigen (HBeAg) positive and hepatitis B e antibody (HBeAb) negative status at screening
* alanine aminotransferase (ALT) ≤ 10 * upper limit of normal (ULN) at screening
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study (and for up to 6 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized
* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal. Post menopausal is defined as:
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 72 hours prior to the start of investigational product

Exclusion Criteria:

* Evidence of decompensated cirrhosis
* Coinfection with human immunodeficiency virus, hepatitis C virus , or hepatitis D virus
* Women who are pregnant or breastfeeding
* Sexually active fertile men not using effective birth control if their partners were WOCBP
* Laboratory values out of protocol-specified range

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (56):
- University Of Connecticut Health Center, Farmington, Connecticut, United States
- Australia (2):
  - Local Institution, Concord, New South Wales
  - Local Institution, Randwick, New South Wales
- Local Institution, Porto Alegre Rs, Rio Grande do Sul, Brazil
- Local Institution, Calgary, Alberta, Canada
- Local Institution, Athens, Greece
- Hong Kong (3):
  - Local Institution, Hong Kong, Hong Kong
  - Local Institution, Shatin, New Territories
  - Local Institution, Tai Po
- India (7):
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Ahmedabad
  - Local Institution, Chandigarh
  - Local Institution, Indore
  - Local Institution, Ludhiana
  - Local Institution, New Delhi
  - Local Institution, Vellore
- Local Institution, Jakarta, Indonesia
- Local Institution, Antella, Firenze, Italy
- Malaysia (2):
  - Local Institution, Kota Kinabalu, Sabah
  - Local Institution, Kuala Lumpur
- Philippines (2):
  - Local Institution, Cebu City
  - Local Institution, Manila
- Poland (5):
  - Local Institution, Chorzów
  - Local Institution, Kielce
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Korea (18):
  - Local Institution, Seoul, Dongdaemun-Gu
  - Local Institution, Ulsan, Donggu
  - Local Institution, Ansan-si, Gyeonggi-do
  - Local Institution, Anyang-si, Gyeonggi-do
  - Local Institution, Bucheon-si, Gyeonggi-do
  - Local Institution, Seongnam-si, Gyeonggi-do
  - Local Institution, Suwon, Gyeonggi-do
  - Local Institution, Koyang, Ilsanseo Gu
  - Local Institution, Incheon, Jung-Gu
  - Local Institution, Seoul, Nowon-Gu
  - Local Institution, Chuncheon
  - Local Institution, Daegu
  - Local Institution, Gangneung
  - Local Institution, Incheon
  - Local Institution, Pusan
  - Local Institution, Seoul
  - Local Institution, Suwon
  - Local Institution, Yangsan
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Tainan R.o.c.
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Chiang Mai
- Turkey (Türkiye) (2):
  - Local Institution, Bornova Izmir
  - Local Institution, Trabzon

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 629 participants were enrolled at 60 sites.
Pre-assignment Details: Of the 629 participants enrolled, 416 were randomized (195 no longer met study criteria, 9 withdrew consent, and 9 had other reason). One participant randomized to entecavir + adefovir (ADV+LVD) Arm withdrew consent before treatment.
Groups:
- Entecavir + Adefovir (ETV+ADV) Combination Therapy: ETV 1.0 mg + ADV 10 mg; Combination therapy given once daily (QD) for 100 weeks
- Entecavir (ETV) Monotherapy: ETV 1.0 mg; QD, for 100 weeks with an option of adding non-study tenofovir (TDF) at Week 48 at the investigator's discretion, and where permitted by the local health authorities and ethics committees.
- Adefovir + Lamivudine (ADV+LVD) Combination Therapy: ADV 10 mg + LVD 100 mg; Combination therapy given QD for 100 weeks
Period: On-Treatment
Arm/Group | Entecavir + Adefovir (ETV+ADV) Combination Therapy | Entecavir (ETV) Monotherapy | Adefovir + Lamivudine (ADV+LVD) Combination Therapy
Started | 138 | 140 | 137
Discontinued Prior to Week 48 Visit | 4 | 2 | 2
Discontinued at or After Week 48 Visit | 2 | 6 | 3
Completed | 63 (Completed the 100 week dosing) | 61 (Completed the 100 week dosing) | 66 (Completed the 100 week dosing)
Not Completed | 75 | 79 | 71
Not completed — Continuing treatment | 69 | 71 | 66
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Other Reason | 0 | 0 | 1
Period: Off-treatment Follow up
Arm/Group | Entecavir + Adefovir (ETV+ADV) Combination Therapy | Entecavir (ETV) Monotherapy | Adefovir + Lamivudine (ADV+LVD) Combination Therapy
Started | 15 | 8 | 14
Completed | 1 | 0 | 2
Not Completed | 14 | 8 | 12
Not completed — Continuing off-treatment follow up | 10 | 8 | 11
Not completed — Follow up not required per protocol | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir + Adefovir (ETV+ADV) Combination Therapy | Entecavir (ETV) Monotherapy | Adefovir + Lamivudine (ADV+LVD) Combination Therapy | Total
Number analyzed (Participants) | 138 | 140 | 137 | 415
Age Continuous [Median (Full Range); unit: years] | 46.0 [18 to 69] | 43.5 [19 to 71] | 43.0 [16 to 74] | 45.0 [16 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 40 | 139
  Male | 91 | 88 | 97 | 276
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 132 | 131 | 126 | 389
  White | 6 | 9 | 11 | 26
Region of Enrollment [Number; unit: participants]
  Australia | 0 | 1 | 1 | 2
  Canada | 1 | 0 | 0 | 1
  Hong Kong | 5 | 7 | 5 | 17
  India | 4 | 3 | 5 | 12
  Indonesia | 0 | 1 | 0 | 1
  Italy | 1 | 0 | 0 | 1
  Korea, Republic of | 108 | 105 | 102 | 315
  Malaysia | 3 | 0 | 2 | 5
  Philippines | 0 | 1 | 1 | 2
  Poland | 5 | 9 | 9 | 23
  Russian Federation | 0 | 0 | 2 | 2
  Singapore | 1 | 1 | 0 | 2
  Taiwan | 8 | 9 | 9 | 26
  Thailand | 1 | 3 | 1 | 5
  Turkey | 1 | 0 | 0 | 1
Hepatitis B surface antigen (HBsAg) status at baseline [Number; unit: participants]
  Positive | 138 | 140 | 137 | 415
  Negative | 0 | 0 | 0 | 0
Hepatitis B e antigen (HBeAg) status at baseline [Number; unit: participants]
  Positive | 138 | 139 | 135 | 412
  Negative | 0 | 1 | 2 | 3
Hepatitis B e antibody (HBeAb) at baseline [Number; unit: participants]
  Positive | 0 | 1 | 2 | 3
  Negative | 138 | 139 | 135 | 412
Alanine Aminotransferase (ALT) [Median (Full Range); unit: U/L] | 49 [10 to 480] | 50 [12 to 367] | 45 [14 to 1300] | 47 [10 to 1300]
LVD-Resistance Substitution [Number; unit: participants] — LVD resistance (LVDr) substitution at reverse transcription codon 204 (M240V/I/S). The participants who did not have LVDr substitution mutations at baseline (day 1) were distributed equally among the 3 study groups (2 with ETV+ADV combination therapy and 3 each with ETV monotherapy and ADV+LVD combination therapy).
  participants
    Present | 136 | 137 | 134 | 407
    Absent | 2 | 3 | 3 | 8
log10 HBV DNA by PCR [Median (Full Range); unit: IU/mL] | 7.6 [4.2 to 9.5] | 7.5 [3.0 to 9.7] | 7.6 [3.2 to 10.0] | 7.6 [3.0 to 10.0]
International Normalization Ratio [Median (Full Range); unit: ratio] | 1.07 [0.80 to 1.97] | 1.07 [0.87 to 2.48] | 1.05 [0.82 to 7.24] | 1.07 [0.80 to 7.24]
Albumin [Median (Full Range); unit: g/dL] | 4.4 [3.1 to 5.1] | 4.5 [3.5 to 5.1] | 4.5 [3.5 to 5.1] | 4.5 [3.1 to 5.1]
Total Bilirubin [Median (Full Range); unit: mg/dL] | 0.6 [0.2 to 1.8] | 0.6 [0.2 to 2.4] | 0.6 [0.2 to 2.6] | 0.6 [0.2 to 2.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) < 50 IU/mL (Approximately 300 Copies/mL) by Polymerase Chain Reaction (PCR) at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan High Pure System (HPS) assay. HBV DNA less than (<)50 International units per milliliter (IU/mL) = approximately 300 copies/mL. Percentage of participants calculated n/N; n= number of participants with HBV DNA <50 IU/mL; N = number of participants analyzed.
Time Frame: Week 48
Population: Participants who received at least 1 dose of study therapy. Participants with missing efficacy assessments were considered as a failure.
Measure: Number; unit: percentage of participants
Groups:
- ETV+ADV Combination Therapy: ETV 1.0 mg + ADV 10 mg; once daily (QD) for 100 weeks
- ETV Monotherapy: ETV 1.0 mg; QD, for 100 weeks with an option of adding non-study tenofovir (TDF) at Week 48 at the investigator's discretion, and where permitted by the local health authorities and ethics committees.
- ADV+LVD Combination Therapy: ADV 10 mg + LVD 100 mg; QD for 100 weeks
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 25.4 | 16.4 | 19.7
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; p = 0.1336, Hochberg procedure; Difference Estimate = 8.9, 95% CI 2-sided [-2.0 to 19.9]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; p = 0.2619, Hochberg procedure; Difference Estimate = 5.7, 95% CI 2-sided [-4.2 to 15.5]

2. Secondary Outcome: Percentage of Participants With HBV DNA < 50 IU/mL (Approximately 300 Copies/mL) by PCR at Week 96
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan HPS assay. HBV DNA < 50 IU/mL = approximately 300 copies/mL. Percentage n/N: n= number of participants with HBV DNA <50 IU/mL; N = number of participants analyzed.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
Percentage of participants | 43.5 | 39.3 | 28.5
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; p = 0.0095, Hochberg procedure; Difference estimate = 15.0, 95% CI 2-sided [3.7 to 26.4]

3. Secondary Outcome: Percentage of Participants Who Achieve HBV DNA < Lower Limit of Quantitation (LOQ = 29 IU/mL [Approximately 169 Copies/mL]) at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan HPS assay. LOQ is the level above which quantitative results may be obtained with a specified degree of confidence. The LOQ is mathematically defined as equal to 10 times the standard deviation of the results for a series of replicates used to determine a justifiable limit of detection. Percentage n/N: n= number of participants with outcome result; N = number of participants analyzed.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 25.4 | 13.6 | 16.8
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 11.8, 95% CI 2-sided [2.5 to 21.1]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 8.6, 95% CI 2-sided [-1.1 to 18.2]

4. Secondary Outcome: Percentage of Participants Who Achieve HBV DNA < Lower Limit of Quantitation (LOQ = 29 IU/mL [Approximately 169 Copies/mL]) at Week 96
Description: as for outcome 3
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
Percentage of participants | 38.4 | 36.4 | 25.5
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference estimate = 12.9, 95% CI 2-sided [1.8 to 23.9]

5. Secondary Outcome: Percentage of Participants Who Achieve HBV DNA < Lower Limit of Detection (LOD = 10 IU/mL [Approximately 58 Copies/mL]) at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan HPS assay. LOD is the lowest concentration level that can be determined to be statistically different from a blank (99% confidence). The LOD is typically determined to be in the region where the signal to noise ratio is greater than 5. Limits of detection are matrix-, method-, and analyte-specific.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 20.3 | 11.4 | 11.7
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 8.9, 95% CI 2-sided [0.3 to 17.4]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 8.6, 95% CI 2-sided [-0.1 to 17.3]

6. Secondary Outcome: Percentage of Participants Who Achieve HBV DNA < Lower Limit of Detection (LOD = 10 IU/mL [Approximately 58 Copies/mL]) at Week 96
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan HPS assay. LOD is the lowest amount or concentration of analyte in a sample, which can be reliably detected, but not necessarily quantified.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 33.3 | 27.1 | 20.4
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference estimate = 12.9, 95% CI 2-sided [2.4 to 23.4]

7. Secondary Outcome: Percentage of Participants With HBV DNA by PCR Category at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan High Pure System (HPS) assay.
Time Frame: Week 48
Population: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants
  < LOQ (29 IU/mL) | 25.4 | 13.6 | 16.8
  LOQ to < 50 | 0 | 2.9 | 2.9
  50 to < 172 | 8.0 | 2.9 | 5.8
  172 to < 1,720 | 26.1 | 7.9 | 12.4
  1,720 to < 17,200 | 28.3 | 22.1 | 31.4
  17,200 to < 172,000 | 8.0 | 25.7 | 24.8
  >= 172,000 | 0.7 | 23.6 | 4.4
  Missing | 3.6 | 1.4 | 1.5

8. Secondary Outcome: Percentage of Participants With HBV DNA by PCR Category at Week 96
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan HPS assay.
Time Frame: Week 96
Population: Participants who received at least 1 dose of study therapy were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants
  < LOQ (29 IU/mL) | 38.4 | 36.4 | 25.5
  LOQ to < 50 | 5.1 | 2.9 | 2.9
  50 to < 172 | 10.1 | 3.6 | 5.8
  172 to < 1,720 | 15.2 | 6.4 | 18.2
  1,720 to < 17,200 | 20.3 | 10.0 | 24.8
  17,200 to < 172,000 | 5.8 | 15.7 | 13.9
  >= 172,000 | 0 | 16.4 | 2.9
  Missing | 5.1 | 8.6 | 5.8

9. Secondary Outcome: Change in Mean log10 From Baseline in HBV DNA at Week 48
Description: HBV DNA was analyzed by PCR, using the Roche COBAS®TaqMan TaqMan HPS assay. Reduction in log10 HBV count=reduced viral load, negative values means reduction.
Time Frame: Baseline, Week 48
Population: Participants who received at least 1 dose of study therapy and had both baseline and post-baseline values. n=participants with baseline and Week 48 values.
Measure: Mean (Standard Error); unit: log10 (IU/mL
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 133 | 138 | 135
log10 (IU/mL
  HBV DNA at Week 48 | 2.79 (0.093) | 4.01 (0.128) | 3.36 (0.111)
  Change from baseline | -4.65 (0.077) | -3.35 (0.117) | -4.11 (0.108)
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Regression, Linear; Difference Estimate = -1.26, 95% CI 2-sided [-1.534 to -0.994]
Statistical Analysis 2: Comparison: ETV Monotherapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Regression, Linear; Difference Estimate = -0.55, 95% CI 2-sided [-0.824 to -0.281]

10. Secondary Outcome: Change in Mean log10 From Baseline in HBV DNA at Week 96
Description: HBV DNA was analyzed by PCR, using the Roche COBAS® TaqMan HPS assay. Reduction in log10 HBV count=reduced viral load.
Time Frame: Baseline, Week 96
Population: Participants who received at least 1 dose of study therapy and had both baseline and post-baseline values were analyzed. n= participants with baseline and Week 96 values.
Measure: Mean (Standard Error); unit: participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 131 | 128 | 129
participants | -5.06 (0.090) | -4.17 (0.163) | -4.49 (0.116)

11. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) > 1 x Upper Limit of Normal (ULN) at Baseline Who Achieve ALT Normalization at Week 48
Description: ALT normalization=ALT level being less than or equal to 1 times the upper limit of normal (ULN). ULN for ALT is 37 or 48 U/L.
Time Frame: Week 48
Population: Participants who received at least 1 dose of study therapy and had ALT > 1 x ULN at baseline (day 1). Participants with missing efficacy assessments were considered as a failure.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 78 | 82 | 69
percentage of participants | 75.6 | 78.0 | 76.8
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = -2.4, 95% CI 2-sided [-15.5 to 10.7]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = -1.2, 95% CI 2-sided [-15.0 to 12.6]

12. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) > 1 x Upper Limit of Normal (ULN) at Baseline Who Achieve ALT Normalization at Week 96
Description: ALT normalization=ALT level being less than or equal to 1 times the upper limit of normal (ULN). ULN for ALT is 37 U/L.
Time Frame: Baseline, Week 96
Population: Participants who received at least 1 dose of study therapy and had ALT > 1 x ULN at baseline (day 1) were analyzed. Participants with missing efficacy assessments were considered as a failure.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 78 | 82 | 69
percentage of participants | 76.9 | 74.4 | 79.7
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = -2.8, 95% CI 2-sided [-16.2 to 10.6]

13. Secondary Outcome: Percentage of Participants With Confirmed HBeAg Loss at Week 48 (Treated HBeAg Positive Participants Only)
Description: HBeAg is a hepatitis B viral protein. HBeAg loss = HBeAg-negative at the specified analysis week
Time Frame: Week 48
Population: Participants who received at least 1 dose of study therapy and were HBeAG positive. Participants with missing efficacy assessments were considered as a failure.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 139 | 135
percentage of participants | 7.2 | 6.5 | 5.9
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 0.8, 95% CI 2-sided [-5.2 to 6.7]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 1.3, 95% CI 2-sided [-4.6 to 7.2]

14. Secondary Outcome: Percentage of Participants With Confirmed HBeAg Loss at Week 96 (Treated HBeAg Positive Participants Only)
Description: HBeAg is a hepatitis B viral protein. HBeAg loss = HBeAg-negative at the specified analysis week
Time Frame: Week 96
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 12.3 | 10.7 | 13.9
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = -1.5, 95% CI 2-sided [-9.5 to 6.4]

15. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 48 (Treated HBeAg-positive Participants Only)
Description: HBeAg is a hepatitis B viral protein. It is an indicator of active viral replication. HBeAg Seroconversion = HBeAg Loss and Presence of Hepatitis B e Antibody (HBeAb).
Time Frame: Week 48
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 139 | 135
percentage of participants | 5.1 | 2.9 | 3.7
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 2.2, 95% CI 2-sided [-2.4 to 6.8]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 1.4, 95% CI 2-sided [-3.5 to 6.2]

16. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 96 (Treated HBeAg-positive Participants Only)
Description: as for outcome 15
Time Frame: Week 96
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 7.2 | 3.6 | 5.1
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 2.1, 95% CI 2-sided [-3.6 to 7.8]

17. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 48
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBsAg loss = HBsAg-negative at the specified analysis week.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 0.7 | 0 | 0.7
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 0.7, 95% CI 2-sided [-0.7 to 2.1]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = -0.0, 95% CI 2-sided [-2.0 to 2.0]

18. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 96
Description: as for outcome 17
Time Frame: Week 96
Population: Participants who received at least 1 dose of study therapy were analyzed. Participants with missing efficacy assessments were considered as a failure.
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 48
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBs seroconversion is defined as HBsAg loss with positive HBsAb.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 0.7 | 0 | 0
Statistical Analysis 1: Comparison: ETV+ADV Combination Therapy vs ETV Monotherapy; Test type: Superiority or Other; Difference Estimate = 0.7, 95% CI 2-sided [-0.7 to 2.1]
Statistical Analysis 2: Comparison: ETV+ADV Combination Therapy vs ADV+LVD Combination Therapy; Test type: Superiority or Other; Difference Estimate = 0.7, 95% CI 2-sided [-0.7 to 2.1]

20. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 96
Description: as for outcome 19
Time Frame: Week 96
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
percentage of participants | 0 | 0 | 0

21. Secondary Outcome: Cumulative Probability of Emergent Genotypic Resistance at Year 1
Description: yr=year. Cumulative probability (CP): Ptotal=1-(1-Pyr1)*(1-Pyr2) where Pyear(i)= number of participants with events at Year i divided by number of participants at risk at Year i for i = 1,2. An "event" is defined as resistance or resistance with virologic breakthrough in a yearly interval. Participants 'at risk' are those who were treated during Year i and did not develop that resistance or resistance with virologic breakthrough prior to Year i. CP were calculated separately for ETV, ADV and TDF resistance. Participants who discontinue from study drug in Year i were assumed to be in follow up for the entire year. (VBT; a ≥ 1 log10 increase in HBV DNA from the on-treatment nadir, confirmed by 2 sequential HBV DNA results or observed at the last on-treatment HBV DNA). ETVr = ETV resistance (rtM204V/I/S plus any substitution at rtT184, rtS202, or rtM250); ADVr/TDFr = ADV/TDF resistance (rtA181T/V or rtN236T = ADVr and TDFr, rtA194T = TDFr only).
Time Frame: Year 1
Population: Treated participants who were tested for resistance, ie. met the following selection criteria. 1) participants with HBV DNA ≥ 50 IU/mL at Week 48 or at the last on-treatment visit and 2) who developed VBT . n=participants
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 139 | 137
percentage of participants
  ETVr : n=134, 134, 134 | 0 | 3 | 0.7
  ADVr /TDFr : n=137, 137, 135 | 0.7 | 0.7 | 1.5
  ETVr or TDFr/ADVr : n=133, 132, 132 | 0.8 | 3.8 | 2.3
  ETVr and TDFr/ADVr : n=138, 139, 137 | 0 | 0 | 0
  ETVr with VBT: n=134, 134, 134 | 0 | 0.7 | 0
  ADVr /TDFr with VBT: n=137, 137, 135 | 0 | 0 | 0
  ETVr or ADVr/TDFr with VBT: n=133, 132, 132 | 0 | 0.8 | 0
  ETVr and ADVr/TDFr with VBT: n=138, 139, 137 | 0 | 0 | 0

22. Secondary Outcome: Cumulative Probability of Emergent Genotypic Resistance at Year 2
Description: Cumulative probability (CP): Ptotal=1-(1-Pyr1)*(1-Pyr2) where Pyear(i)= number of participants with events at Year i divided by number of participants at risk at Year i for i = 1,2. An "event" is defined as resistance or resistance with virologic breakthrough in a yearly interval. Participants 'at risk' are those who were treated during Year i and did not develop that resistance or resistance with virologic breakthrough prior to Year i. CP were calculated separately for ETV, ADV and TDF resistance. Participants who discontinue from study drug in Year i were assumed to be in follow up for the entire year. (VBT; a ≥ 1 log10 increase in HBV DNA from the on-treatment nadir, confirmed by 2 sequential HBV DNA results or observed at the last on-treatment HBV DNA). ETVr = ETV resistance (rtM204V/I/S plus any substitution at rtT184, rtS202, or rtM250); ADVr/TDFr = ADV/TDF resistance (rtA181T/V or rtN236T = ADVr and TDFr, rtA194T = TDFr only).
Time Frame: Year 2
Population: Treated participants who were tested for resistance were analyzed, ie. They met the following selection criteria: 1) participants with HBV DNA ≥ 50 IU/mL at Week 96 or at the last on-treatment visit and 2) who developed VBT. n=participants
Measure: Number; unit: percentage of participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 134 | 137 | 135
percentage of participants
  ETVr : n=130, 128, 131 | 0.8 | 9.8 | 1.5
  ADVr/TDFr : n=132, 134, 131 | 0.7 | 1.5 | 2.2
  ETVr or ADVr/TDFr : n=128, 125, 127 | 1.5 | 10.7 | 3.8
  ETVr and ADVr/TDFr : n=134, 137, 135 | 0 | 0.7 | 0
  ETVr with VBT: n=130, 128, 131 | 0 | 6.2 | 0
  ADVr/TDFr with VBT: n=132, 134, 131 | 0 | 0.7 | 0
  ETVr or ADVr/TDFr with VBT: n=128, 125, 127 | 0 | 6.3 | 0
  ETVr and ADVr/TDFr with VBT: n=134, 137, 135 | 0 | 0.7 | 0

23. Secondary Outcome: Participants With Adverse Events (AE), Serious Adverse Events (SAE), and Discontinuations Due to Adverse Events or Laboratory Abnormalities During Treatment
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded. Grade 1 = mild, Grade 2= moderate, Grade 3 = severe, Grade 4 = life threatening/disabling, Grade 5 = death.
Time Frame: From start of study therapy through Week 100 + 5 days
Population: All treated participants.
Measure: Number; unit: participants
Groups:
- ETV+ADV Combination Therapy: ETV 1.0 mg + ADV 10 mg; QD for 100 weeks
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
participants
  Deaths | 0 | 0 | 1
  SAEs | 11 | 17 | 12
  Discontinuations due to AEs | 1 | 2 | 2
  AEs | 101 | 109 | 92
  Grade 2-4 Related AEs | 2 | 12 | 1
  Grade 3-4 Related AEs | 5 | 7 | 9

24. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Hematology
Description: Criteria for hematology abnormalities were: Hemoglobin: <=11.0 g/dL; White Blood Cells: <4000/mm^3; Absolute Neutrophils (includes absolute bands): <1500/mm^3; Platelets: <=99,000/mm^3; International Normalized Ratio: ≥ 1.5 and ≥ 0.5 from baseline.
Time Frame: From start of study through Week 100 + 5 days
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
participants
  Hemoglobin | 8 | 9 | 11
  White Blood Cells | 53 | 48 | 38
  Neutrophils | 14 | 17 | 15
  Platelets | 13 | 14 | 12
  International Normalized Ratio | 8 | 7 | 9

25. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Serum Chemistry
Description: ULN=upper limit of normal (Normal ranges are Central lab data and vary according to the site). ALT:>1.25*ULN, AST:>1.25*ULN, ALP:>1.25*ULN, Total Bilirubin:>1.1*ULN, Serum Lipase:>1.10*ULN, Creatinine:>1.1*ULN, Blood Urea Nitrogen:1.25*ULN, Hyperglycemia:>116 mg/dL, Hypoglycemia:<64 mg/dL, Hyponatremia:<132meq/L, Hypokalemia:<3.4 meq/L, Albumin:≥1g/dL decrease from baseline, <3 g/dL; Hypernatremia:>148 meq/L, Hyperkalemia:>5.6 meq/L, Hypokalemia:<3.4 meq/L, Hyperchloremia:>113 meq/L, Hypochloremia:<93 meq/L; ALT flare: on treatment (OT), >2*Baseline and >10*ULN; off treatment (OF), 2*end of dosing value and >10*ULN
Time Frame: On treatment : Day 1 through Week 100 + 5 days; Offtreatment = End of OT period through 24 weeks
Population: All treated participants. n = number of participants in the OF period.
Measure: Number; unit: participants
Arm/Group | ETV+ADV Combination Therapy | ETV Monotherapy | ADV+LVD Combination Therapy
Number analyzed (Participants) | 138 | 140 | 137
participants
  Alanine aminotransferase (ALT) | 76 | 83 | 74
  Aspartate aminotransferase (AST) | 60 | 62 | 53
  Alkaline Phosphatase (ALP) | 8 | 4 | 6
  Albumin | 1 | 1 | 1
  Serum Lipase | 24 | 33 | 24
  Creatinine | 2 | 2 | 4
  Blood Urea Nitrogen | 0 | 1 | 2
  Hyperglycemia | 39 | 46 | 37
  Hypoglycemia | 9 | 5 | 9
  Hypernatremia | 10 | 10 | 10
  Hyponatremia | 0 | 0 | 0
  Hyperkalemia | 3 | 4 | 5
  Hypokalemia | 4 | 2 | 2
  Hyperchloremia | 1 | 1 | 1
  Hypochloremia | 1 | 0 | 0
  ALT flare - Ontreatment | 3 | 2 | 2
  ALT flare - Offtreatment | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 96
Groups:
- ADV + LVD Combination Therapy: ADV 10 mg + LVD 100 mg; QD for 100 weeks
- ETV + ADV Combination Therapy: ETV 1.0 mg + ADV 10 mg; once daily (QD) for 100 weeks
Arm/Group | ADV + LVD Combination Therapy | ETV Monotherapy | ETV + ADV Combination Therapy
Serious Adverse Events (participants affected / at risk) | 13/137 | 21/140 | 14/138
Other Adverse Events (participants affected / at risk) | 62/137 | 75/140 | 63/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADV + LVD Combination Therapy (N=137) | ETV Monotherapy (N=140) | ETV + ADV Combination Therapy (N=138)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Intracranial hypotension (Nervous system disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0
Optic atrophy (Eye disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 4
Hydrocephalus (Nervous system disorders) | 1 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADV + LVD Combination Therapy (N=137) | ETV Monotherapy (N=140) | ETV + ADV Combination Therapy (N=138)
Hepatic steatosis (Hepatobiliary disorders) | 9 | 8 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 7 | 5
Headache (Nervous system disorders) | 13 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 19 | 28 | 23
Abdominal pain upper (Gastrointestinal disorders) | 6 | 10 | 5
Hypertension (Vascular disorders) | 3 | 7 | 2
Abdominal discomfort (Gastrointestinal disorders) | 7 | 3 | 8
Alanine aminotransferase increased (Investigations) | 5 | 8 | 8
Nausea (Gastrointestinal disorders) | 4 | 8 | 6
Dyspepsia (Gastrointestinal disorders) | 8 | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 2
Fatigue (General disorders) | 8 | 4 | 4
Nasopharyngitis (Infections and infestations) | 8 | 17 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.